CLINICAL TRIAL: NCT01136837
Title: The Prognostic Significance of a Fragmented QRS Complex After Primary Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Hasan Arı, Bursa Postgraduate Hospital
Other Study IDs: BYİEAH-3
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2008-11

CONDITIONS: Fragmented QRS; Primary PCI; MACE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fragmented QRS positive: fQRS at 48 hours after Primary PCI
  Interventions: Other: primary pcı

INTERVENTIONS:
Other: primary pcı

SUMMARY:
To investigate the prognostic significance of a fragmented QRS (fQRS) complex in a patient who had undergone primary percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain that continued longer than 30 minutes and with ≥ 2 mm ST elevation in ECG at least in two adjacent derivations were diagnosed with an acute STEMI. In all patients, at least two-fold increases were seen in serum CK-MB levels compared to normal values.Having acute STEMI for the first time was stipulated for inclusion in the study.

Exclusion Criteria:

* Subjects with known allergies to aspirin and clopidogrel, inadequate echocardiographic images, malignancy, a previous cerebrovascular event, renal dysfunction (creatine level > 2.5 mg/dl), a previous MI, or a history of cardiogenic shock as well as those who refused to participate in the study were excluded.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who presented to the hospital within 12 hours of the onset of chest pain who were admitted to the coronary intensive care unit (ICU) with the diagnosis of acute STEMI and who were administered primary PCI. Having acute STEMI for the first time was stipulated for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events
  the presence of a fQRS at 48 hours after primary PCI is a significant parameter in predicting adverse cardiovascular events;

SECONDARY OUTCOMES:
Q Wave and QRS distortion for predicting major adverse cardiac events
  the presence of a fQRS is a more sensitive and specific parameter in predicting development of adverse cardiovascular events than Q wave and QRS distortion; and compared to Q wave, fQRS correlated more significantly with the presence of a scar

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Bursa, Turkey (Türkiye)

REFERENCES:
- [Derived] Ari H, Cetinkaya S, Ari S, Koca V, Bozat T. The prognostic significance of a fragmented QRS complex after primary percutaneous coronary intervention. Heart Vessels. 2012 Jan;27(1):20-8. doi: 10.1007/s00380-011-0121-9. Epub 2011 Feb 23. PMID 21344317